CLINICAL TRIAL: NCT03901404
Title: Used During Myomectomy Operation; Comparison of Fundus Incision, Energy Modalities and Methods of Extraction
Brief Title: Myomectomy Operation and Fundus Incision, Energy Modalities and Methods of Extraction
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and GynecologyR, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.12.67
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Myoma;Uterus; Surgery
Keywords: Myomectomy; Fundus Incision; Energy Modalities; Methods of Extraction
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Myomectomy Operation — Patients undergoing myomectomy for myoma uteri

SUMMARY:
Myomectomy operation due to myoma uteri is an operation that can cause serious blood loss. For some anatomical reasons, fundal myomas were removed, while a group of investigators recommended the initiation of a longitudinal incision and some surgeons preferred a transverse incision. the authors aim to show some surgical differences, intraoperative blood loss, and difficulties and ease of removal of myoma in patients with these approaches without consensus. It is also noted that the incision made with the same energy modality is recorded; The effect of energy modality on blood loss and surgical comfort will be examined. Different approaches are used for laparoscopic surgical operations in order to remove myoma from the abdomen. It can be removed from the vagina by colpotomy and can also be minimized in the abdomen by a morselator. In particular, patients with vaginal myoma removed, such as complaints of postoperative dyspareunia will be followed. In this way, the investigators aim to evaluate the methods which have not yet gained clarity in the literature or have not proven superiority to each other.

ELIGIBILITY:
Inclusion Criteria:

- Patients operated with the diagnosis of myoma uteri

Exclusion Criteria:

* Cardiopulmonary diseases such as cardiac insufficiency, myocardial infarction, unstable angina, acute or new vascular thrombosis, asthma or pulmonary obstructive disease;
* Patients with long-term Trendelenburg contraindications;
* Previous pelvic or abdominal radiation therapy; or those with inadequate bone marrow, kidney and hepatic function;
* Gynecological malignancies.
* Those who received preoperative medication due to myoma uteri

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients operated with the diagnosis of myoma uteri
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Fundus Incision | 3 months
  In patients undergoing myomectomy, the incision used by the surgeon will be recorded to remove myoma. to be recorded as transverse or vertical.
Energy Modalities | 3 months
  In patients undergoing myomectomy, the energy modality used by the surgeon will be recorded to remove the myoma.
  bipolari, monopolar or ultrasonic
Methods of Extraction | 3 months
  In patients undergoing myomectomy operation, the method used by the surgeon to remove myoma from the abdomen will be recorded.
  morselator, vaginally with colpotomi

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)